CLINICAL TRIAL: NCT06645704
Title: An Open-Label Phase 1 Study in Healthy Male Subjects to Investigate the Absorption, Metabolism and Excretion of [14C]-EP262 Following Single-Dose Oral Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Escient Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP-262-104
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-EP262 25 mg (Experimental): Administered orally.
  Interventions: Drug: EP262

INTERVENTIONS:
Drug: EP262 — Single dose of [14C]-EP262 administered orally.

SUMMARY:
This study is being conducted to assess the mass balance, pharmacokinetics, and metabolite profiles of a single oral dose of [14C]-EP262 in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18 to 55 years
* Body mass index of 18 to 32 kg/m2 and body weight of 55 to 100 kg
* Negative result for HIV, HBV, and HCV at Screening
* Male subjects with female partners of reproductive potential must be surgically sterile or use adequate birth control
* No use of tobacco or nicotine containing products within the past 6 months

Exclusion Criteria:

* History or presence of any condition or prior surgery that could pose a significant risk in the opinion of the investigator
* History of malignancy within the past 5 years
* History of any serious allergic reactions or hypersensitivity
* Recent history of incomplete bladder emptying with voiding or awakening more than once at a night to void
* Usual habit of bowel movements of less than 1 or more than 3 bowel movements per day

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Mass balance of [14C]-EP262 | Measured from Day 1 to End of Study or Early Termination (Approximately 1 month)
  Assessed by the total recovery of radioactivity from urine and feces
Pharmacokinetics (PK) of EP262 and [14C] | Measured from Day 1 to End of Study or Early Termination (Approximately 1 month)
  Assessed by the concentration of EP262 in plasma and [14C] in whole blood, plasma, urine, and feces

SECONDARY OUTCOMES:
Metabolite profile of EP262 | Measured from Day 1 to End of Study or Early Termination (Approximately 1 month)
  Assessed by the concentration of EP262 metabolites in plasma, urine, and feces
Safety and tolerability of [14C]-EP262 | Measured from Day 1 to End of Study or Early Termination (Approximately 1 month)
  Assessed by the incidence of treatment emergent adverse events, clinical laboratory evaluations, vital signs, 12-lead electrocardiogram, and physical examination findings

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron Clinical Pharmacology Center (CPC), Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No